CLINICAL TRIAL: NCT05425550
Title: Evaluation of the Medidux™ Digital Health Application in Patients With HER2-positive Breast Cancer During Chemotherapy in Combination With HER2-targeted Therapy (Including Tyrosine Kinase Inhibitors [TKI]) or an Antibody-drug Conjugate Therapy: a Multicenter Randomized Controlled Trial.
Brief Title: Evaluation of the Medidux™ Digital Health Application in Patients With HER2-positive Breast Cancer.
Acronym: PRO2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was discontinued due to low recruitment rates. Despite various measures, such as training courses and workshops, recruitment rates could not be improved in the long term.
Sponsor: Palleos Healthcare GmbH (Industry)
Collaborators: Mobile Health AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO2
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: app; PRO2; medidux; ePro; palleos; xlife science; mobile Health AG; mobile Health; medical device; palleos healthcare
MeSH Terms: conditions — Breast Neoplasms; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Experimental group is using the medidux™ app
  Interventions: Device: medidux™ app
- Arm B (No Intervention): Control group does not use the medidux™ app

INTERVENTIONS:
Device: medidux™ app — Use of the regular medidux™ application for 12 (maximum 16) weeks
  Arms: Arm A

SUMMARY:
Multicenter, prospective, randomised and controlled study to evaluate the medidux™ app during an observation period of 12 weeks (maximum 16 weeks in case of shifts in the initially planned therapy).

DETAILED DESCRIPTION:
The PRO2 study is being conducted by palleos healthcare GmbH, the sponsor of the study, with the participation of an expected 585 patients at 40 study sites in Germany and 10 study sites in the German-speaking part of Switzerland with the aim of investigating the medical benefit of the smartphone application medidux™ (app) with regard to the occurrence of side effects in breast cancer therapy. Furthermore, the potential impact on the application of the chemotherapy or antibody-drug conjugate, respectively, the number of unplanned doctor visits, as well as hospitalizations and how often the app is used will be investigated.

The app was developed by mobile Health AG and is intended to accompany therapy. It is an approved CE-marked medical device that will be used in the study within the intended purpose. Study participants can use the app to document symptoms and well-being, as well as vital signs (e.g., blood pressure), and complete a test that can be used to assess mental performance. The entries can be viewed by the study physician through the medidux™ web application. The study participants can refer to the entries during the treatment visit to explain the course of therapy and perceived symptoms. As part of the study, use of the app will be compared to the normal treatment routine (without the app). A randomization process will determine whether study participants receive the app. The probability of receiving the app is 50%. If study participants receive the app, it can be used after installation on the personal smartphone. The approximately 12- to a maximum of 16-week observation period begins with the regular breast cancer therapy. The specific treatment of the breast cancer is not interfered with during the study, i.e. the administration of the therapy itself is carried out in the same way as it would be without the app.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with signed informed consent.
2. Female and male patients, age at diagnosis 18 years and older.
3. Patients with HER2-positive breast carcinoma* (confirmed by a local pathologist).
4. Patients with breast carcinoma with positive or negative hormone receptor status.
5. Patients prior to initiation of neoadjuvant, adjuvant or palliative chemotherapy** in combination with HER2-targeted therapy (including tyrosine kinase inhibitors [TKI]) or an antibody-drug conjugate therapy.
6. ECOG performance Status ≤ 1.
7. Sufficient command of the German language as assessed by the investigator.
8. Presence of a personal smartphone with iOS or Android system. The operating system must be updated to the latest, second or third most recent major version and the medidux™ app must be installed prior to the start of the first treatment cycle.

   * * HER2-positive in the context of the study defined as "eligible for an approved HER2-targeted therapy," i.e., in addition to immunohistochemistry (IHC) scores of 3+ and 2+ with positive results of in-situ hybridization (ISH+), also according to new standard HER2 low (IHC 1+ and 2+ with simultaneous negative result of in-situ-hybridization (ISH-))
   * ** Patients receiving chemotherapy in combination with HER2-targeted therapy as part of a (neo)adjuvant sequence therapy (e.g. as second part after previous EC therapy) may be included. Accordingly, the PRO2 study will not start until patients begin combination of chemotherapy and HER2-targeted therapy.

Exclusion Criteria:

1. Patients for whom it is questionable whether they will follow the study protocol, e.g., due to psychological problems or their private life situation.
2. Patients with insufficient knowledge about the use of smartphones.
3. Patients at the start of therapy with an ECOG performance status ≥ 2.
4. Patients who have already used the medidux™ app or its predecessor consilium care™ before admission to the study.
5. Patients with breast carcinoma who are to be treated exclusively with HER2-targeted antibody monotherapy or TKI-therapy without simultaneous chemotherapy. The sole administration of antibody-drug conjugates alone is permitted/prescribed by the SmPC.
6. Simultaneous participation in an interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events (AEs) (CTCAE severity >2) and serious AEs (SAE) within the observation period. | From the day of randomization until Day 84; maximum observation period is 16 weeks (112 days)
  As the primary endpoint, the occurrence of adverse events, either of type SAE or of type AE with CTCAE severity >2, with a start date within the observation period will be measured for each patient. In the following, these events are referenced as high-grade AEs (HAE).
  The parameters included in the primary endpoint analysis are recorded by the investigator during regular study visits within 12 weeks. The observation period can, however, be extended to the period required for the completion of the initially planned therapy due to shifts in therapy; the maximum observation period is limited to 16 weeks. Adverse events are mapped to the hierarchy and thesaurus terms of the Medical Dictionary for Regulatory Activities (MedDRA, latest version). Severity will be determined according to NCI CTCAE v5.0.
  In addition to the assessment by the investigators and the medical monitor, the HAEs will be assessed by a blinded medical expert (Adjudicator) and a classification is made independently.

SECONDARY OUTCOMES:
Adverse events (AE) occurring in the observation period recorded and assessed by the investigator during the scheduled study visits. | From the day of randomization until Day 84; maximum observation period is 16 weeks (112 days)
  Adverse events (AE) occurring in the observation period recorded and assessed by the investigator during the scheduled study visits. Events classified as "hair loss" (alopecia) are excluded from the analysis as they cannot be influenced a priori by the medidux™ app but may be subject to a technological center bias due to the availability of "cold caps", which cannot be controlled within the scope of the study. Adverse events are mapped to hierarchy and thesaurus terms of the Medical Dictionary for Regulatory Activities (MedDRA, latest version). Severity is determined according to NCI CTCAE v5.0.
Serious adverse events (SAEs) | From the day of randomization until Day 84; maximum observation period is 16 weeks (112 days)
  Serious adverse events (SAEs), defined as a subset of the adverse events defined under Outcome 2 that are classified as "serious".
Number of patients with at least one documented chemotherapy (CTX) respectively antibody-drug conjugate dose reduction. | From the day of randomization until Day 84; maximum observation period is 16 weeks (112 days)
  Number of patients with at least one documented chemotherapy (CTX) respectively antibody-drug conjugate dose reduction.
CTX respectively antibody-drug conjugate adherence | From the day of randomization until Day 84; maximum observation period is 16 weeks (112 days)
  CTX respectively antibody-drug conjugate adherence defined as the percentage of cumulative chemotherapy respectively antibody-drug conjugate dose actually received relative to the planned cumulative dose.
Number of treatment-associated unplanned emergency consultations | From the day of randomization until Day 84; maximum observation period is 16 weeks (112 days)
  Unplanned emergency consultations are defined as emergency-related consultations outside of planned treatment or follow-up visits to the treatment center or the investigator, as well as unplanned visits to other physicians or emergency services.
Number of hospitalisations | From the day of randomization until Day 84; maximum observation period is 16 weeks (112 days)
  Number of hospitalisations defined as inpatient admission at the center or at another medical facility because of an (S)AE
Number and severity of symptoms recorded by medidux™ in the experimental arm. | From the day of randomization until Day 84; maximum observation period is 16 weeks (112 days)
  Number and severity of symptoms recorded by medidux™ (for ePRO modified NCI CTCAE 4.0 subset of 106 items for cancer) in the experimental arm. ePRO symptoms can be continuously documented via the app by the patient.
Adherence | From the day of randomization until Day 84; maximum observation period is 16 weeks (112 days)
  Adherence defined for the experimental arm as the percentage of days in the observation period on which any form of use of the medidux™ app took place.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Trojan, Prof. Dr., Principal Investigator — Seespital Horgen-Onkologie; Peter Fasching, Prof. Dr., Principal Investigator — Universitätsklinikum Erlangen; Frauenklinik
Locations (1):
- Seespital Horgen-Onkologie, Horgen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emanuel EJ, Wendler D, Grady C. What makes clinical research ethical? JAMA. 2000 May 24-31;283(20):2701-11. doi: 10.1001/jama.283.20.2701. PMID 10819955
- [Background] Gnanasakthy A, DeMuro C, Clark M, Haydysch E, Ma E, Bonthapally V. Patient-Reported Outcomes Labeling for Products Approved by the Office of Hematology and Oncology Products of the US Food and Drug Administration (2010-2014). J Clin Oncol. 2016 Jun 1;34(16):1928-34. doi: 10.1200/JCO.2015.63.6480. Epub 2016 Apr 11. PMID 27069082
- [Background] Bennett AV, Jensen RE, Basch E. Electronic patient-reported outcome systems in oncology clinical practice. CA Cancer J Clin. 2012 Sep-Oct;62(5):337-47. doi: 10.3322/caac.21150. Epub 2012 Jul 18. PMID 22811342
- [Background] Prince RM, Atenafu EG, Krzyzanowska MK. Hospitalizations During Systemic Therapy for Metastatic Lung Cancer: A Systematic Review of Real World vs Clinical Trial Outcomes. JAMA Oncol. 2015 Dec;1(9):1333-9. doi: 10.1001/jamaoncol.2015.3440. PMID 26378774
- [Background] Whitney RL, Bell JF, Tancredi DJ, Romano PS, Bold RJ, Wun T, Joseph JG. Unplanned Hospitalization Among Individuals With Cancer in the Year After Diagnosis. J Oncol Pract. 2019 Jan;15(1):e20-e29. doi: 10.1200/JOP.18.00254. Epub 2018 Dec 5. PMID 30523749
- [Background] Brooks GA, Abrams TA, Meyerhardt JA, Enzinger PC, Sommer K, Dalby CK, Uno H, Jacobson JO, Fuchs CS, Schrag D. Identification of potentially avoidable hospitalizations in patients with GI cancer. J Clin Oncol. 2014 Feb 20;32(6):496-503. doi: 10.1200/JCO.2013.52.4330. Epub 2014 Jan 13. PMID 24419123
- [Background] McKenzie H, Hayes L, White K, Cox K, Fethney J, Boughton M, Dunn J. Chemotherapy outpatients' unplanned presentations to hospital: a retrospective study. Support Care Cancer. 2011 Jul;19(7):963-9. doi: 10.1007/s00520-010-0913-y. Epub 2010 May 25. PMID 20499108
- [Background] Henry DH, Viswanathan HN, Elkin EP, Traina S, Wade S, Cella D. Symptoms and treatment burden associated with cancer treatment: results from a cross-sectional national survey in the U.S. Support Care Cancer. 2008 Jul;16(7):791-801. doi: 10.1007/s00520-007-0380-2. Epub 2008 Jan 17. PMID 18204940
- [Background] Dufton PH, Drosdowsky A, Gerdtz MF, Krishnasamy M. Socio-demographic and disease related characteristics associated with unplanned emergency department visits by cancer patients: a retrospective cohort study. BMC Health Serv Res. 2019 Sep 6;19(1):647. doi: 10.1186/s12913-019-4509-z. PMID 31492185
- [Background] Egbring M, Far E, Roos M, Dietrich M, Brauchbar M, Kullak-Ublick GA, Trojan A. A Mobile App to Stabilize Daily Functional Activity of Breast Cancer Patients in Collaboration With the Physician: A Randomized Controlled Clinical Trial. J Med Internet Res. 2016 Sep 6;18(9):e238. doi: 10.2196/jmir.6414. PMID 27601354
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Background] Trojan A, Huber U, Brauchbar M, Petrausch U. Consilium Smartphone App for Real-World Electronically Captured Patient-Reported Outcome Monitoring in Cancer Patients Undergoing anti-PD-L1-Directed Treatment. Case Rep Oncol. 2020 May 12;13(2):491-496. doi: 10.1159/000507345. eCollection 2020 May-Aug. PMID 32518544
- [Background] Pircher M, Winder T, Trojan A. Response to Vemurafenib in Metastatic Triple-Negative Breast Cancer Harbouring a BRAF V600E Mutation: A Case Report and Electronically Captured Patient-Reported Outcome. Case Rep Oncol. 2021 Mar 29;14(1):616-621. doi: 10.1159/000513905. eCollection 2021 Jan-Apr. PMID 33976643
- [Background] Schmalz O, Jacob C, Ammann J, Liss B, Iivanainen S, Kammermann M, Koivunen J, Klein A, Popescu RA. Digital Monitoring and Management of Patients With Advanced or Metastatic Non-Small Cell Lung Cancer Treated With Cancer Immunotherapy and Its Impact on Quality of Clinical Care: Interview and Survey Study Among Health Care Professionals and Patients. J Med Internet Res. 2020 Dec 21;22(12):e18655. doi: 10.2196/18655. PMID 33346738
- [Background] Trojan A, Battig B, Mannhart M, Seifert B, Brauchbar MN, Egbring M. Effect of Collaborative Review of Electronic Patient-Reported Outcomes for Shared Reporting in Breast Cancer Patients: Descriptive Comparative Study. JMIR Cancer. 2021 Mar 17;7(1):e26950. doi: 10.2196/26950. PMID 33729162
- [Background] Trojan A, Leuthold N, Thomssen C, Rody A, Winder T, Jakob A, Egger C, Held U, Jackisch C. The Effect of Collaborative Reviews of Electronic Patient-Reported Outcomes on the Congruence of Patient- and Clinician-Reported Toxicity in Cancer Patients Receiving Systemic Therapy: Prospective, Multicenter, Observational Clinical Trial. J Med Internet Res. 2021 Aug 5;23(8):e29271. doi: 10.2196/29271. PMID 34383675
- [Background] Carpenter JR, Roger JH, Kenward MG. Analysis of longitudinal trials with protocol deviation: a framework for relevant, accessible assumptions, and inference via multiple imputation. J Biopharm Stat. 2013;23(6):1352-71. doi: 10.1080/10543406.2013.834911. PMID 24138436
- [Background] Hsieh FY, Bloch DA, Larsen MD. A simple method of sample size calculation for linear and logistic regression. Stat Med. 1998 Jul 30;17(14):1623-34. doi: 10.1002/(sici)1097-0258(19980730)17:143.0.co;2-s. PMID 9699234
- [Background] Maansson R, Radley D, Jiang Q, Beeslaar J, Patterson S, Absalon J, Perez J. Modeling excess zeroes in an integrated analysis of vaccine safety. Hum Vaccin Immunother. 2018 Jun 3;14(6):1530-1533. doi: 10.1080/21645515.2018.1433972. Epub 2018 Feb 23. PMID 29393713
- [Background] Zhu H, Lakkis H. Sample size calculation for comparing two negative binomial rates. Stat Med. 2014 Feb 10;33(3):376-87. doi: 10.1002/sim.5947. Epub 2013 Aug 23. PMID 24038204
- [Background] van Buuren S, Groothuis-Oudshoorn K. mice: Multivariate Imputation by Chained Equations in R. Journal of Statistical Software 2011, 45(3), 1-67. doi: 10.18637/jss.v045.i03
- [Derived] Trojan A, Kuhne C, Kiessling M, Schumacher J, Drose S, Singer C, Jackisch C, Thomssen C, Kullak-Ublick GA. Impact of Electronic Patient-Reported Outcomes on Unplanned Consultations and Hospitalizations in Patients With Cancer Undergoing Systemic Therapy: Results of a Patient-Reported Outcome Study Compared With Matched Retrospective Data. JMIR Form Res. 2024 May 6;8:e55917. doi: 10.2196/55917. PMID 38710048
- See also: National Cancer Institute. Common Terminology Criteria for Adverse Events v.4.0 (CTCAE). Accessed March 8th, 2017. — http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm